CLINICAL TRIAL: NCT00938379
Title: Clinical Evaluation of Insect Repellent and Insecticide Treated Nets Against Malaria, JE & Dengue in Rural Communities in Lao PDR
Brief Title: Clinical Evaluation of Insect Repellent and Insecticide Treated Nets in Lao PDR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Population Services International (Other)
Responsible Party: Dr Nigel Hill, Head of Unit, Disease Control & Vector Biology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NHLAO1
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Malaria; Dengue; Japanese Encephalitis
Keywords: mosquito; repellent; vector control; malaria
MeSH Terms: conditions — Malaria; Dengue; Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20% deet insect repellent (Experimental): experimental intervention
  Interventions: Drug: 20% deet insect repellent
- lotion without repellent active (Placebo Comparator)
  Interventions: Drug: placebo control

INTERVENTIONS:
Drug: 20% deet insect repellent — skin-applied repellent lotion
  Arms: 20% deet insect repellent
Drug: placebo control — Identical base formulation of lotion but without any deet active
  Arms: lotion without repellent active

SUMMARY:
Rural communities involved in agriculture are often at highest risk of insect-borne diseases in Southeast (SE) Asia.

Skin-applied insect repellents may prove a useful means of reducing mosquito-borne diseases for those people working outdoors in high risk areas.

This trial is evaluating the use of insect repellent (20% diethyltoluamide) to reduce incidence of malaria, Japanese Encephalitis and Dengue. The investigators will recruit up to 1000 households from 100 villages in rural Laos. In each house the investigators shall recruit up to 5 individuals. Half of households will be randomised to repellent, half to a placebo. All individuals will be provided with insecticide treated bed nets for use at night. All household occupants will be followed for 7 months to record malaria cases by Rapid Diagnostic Test every month. Blood spots will be collected at start and end of study to measure Japanese Encephalitis and Dengue. All positive cases will be promptly treated. Outcome will be reduction in number of malaria cases (primary outcome) and Dengue/Japanese Encephalitis (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* working in agriculture
* available for monthly follow-up

Exclusion Criteria:

* allergy to repellent
* pregnant / breastfeeding

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
reduction in malaria incidence | monthly over 7 months

SECONDARY OUTCOMES:
Reduction in Japanese Encephalitis and / or Dengue infections | After 7 months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hill, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Rural villages in Attepu and Sekong Provinces, Laos PDR, Pakse, Attepu, Laos

REFERENCES:
- [Derived] Chen-Hussey V, Carneiro I, Keomanila H, Gray R, Bannavong S, Phanalasy S, Lindsay SW. Can topical insect repellents reduce malaria? A cluster-randomised controlled trial of the insect repellent N,N-diethyl-m-toluamide (DEET) in Lao PDR. PLoS One. 2013 Aug 14;8(8):e70664. doi: 10.1371/journal.pone.0070664. eCollection 2013. PMID 23967083